CLINICAL TRIAL: NCT02370355
Title: Assessment of Novel Biomarkers in Patients With Metastatic Castration Resistant Prostate Cancer
Brief Title: Molecular Characterization of CTCs and ctDNA in Blood and Plasma Samples From Patients With Metastatic and/or Hormone-Resistant Prostate Cancer
Status: Terminated | Type: Observational
Why Stopped: Sponsor decided not to pursue study
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 4P-14-6; NCI-2014-02682 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HS-14-00861; 4P-14-6 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2015-02-17; First posted 2015-02-24 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Hormone-Resistant Prostate Cancer; Metastatic Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Blood, plasma, and tissue (optional)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I (retrospective analysis): Previously collected plasma samples are analyzed for ctDNA via PCR and NSG.
  Interventions: Other: Laboratory Biomarker Analysis
- Group II (prospective analysis): Patients undergo collection of blood samples before and following systemic therapy for analysis of CTC enumeration, RNA expression, and ctDNA via PCR and NSG.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of blood samples
  Other Names: Cytologic Sampling
  Groups: Group II (prospective analysis)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies molecular characterization of circulating tumor cells (CTCs) and circulating tumor (ct) deoxyribonucleic acid (DNA) in blood and plasma samples from patients with prostate cancer that has spread to other places in the body and/or has not responded to previous treatment with hormones. Studying samples of blood and plasma collected from patients with prostate cancer before, during, and/or after treatment in the laboratory may help doctors learn more about changes that occur in DNA and identify the development of drug resistance.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Perform molecular analysis of plasma samples from 25 patients with metastatic prostate cancer collected before and during treatment of the disease with abiraterone acetate (Zytiga) or enzalutamide (Xtandi).

II. Perform molecular characterization of circulating tumor cells (CTCs) and plasma collected from 75 patients with progressing advanced metastatic prostate cancer.

OUTLINE: Patients are assigned to 1 of 2 groups based on the timing of specimen collection.

GROUP I: Previously collected plasma samples are analyzed for ctDNA via polymerase chain reaction (PCR) and next generation sequencing (NSG).

GROUP II: Patients undergo collection of blood samples before and following systemic therapy for analysis of CTC enumeration, ribonucleic acid (RNA) expression, and ctDNA via PCR and NSG.

ELIGIBILITY:
Inclusion Criteria:

* GROUP I: Samples for Group I will be selected from existing sample sets obtained from concluded studies (USC IRB #'s 10-00006 and 11-00450)
* GROUP I: Excess plasma collected and stored in these trials from patients treated with abiraterone or enzalutamide will be used for the molecular analysis of the current protocol
* GROUP II: The second group of samples (Group 2) will involve prospective collection of peripheral blood from patients with advanced, treatment-resistant metastatic prostate cancer
* GROUP II: Histologic documentation of prostate cancer
* GROUP II: Metastatic cancer diagnosed by imaging and other clinical criteria
* GROUP II: Treatment-resistance determined by at least one of the following factors: increase in prostate-specific antigen (PSA) value over a baseline measurement; increase in size or number of metastatic deposits determined on imaging; and/or progression in cancer related symptoms

Min Age: 19 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic and/or hormone-resistant prostate cancer consented under University of Southern California (USC) protocols IRB numbers 10-00006 and 11-004500 or treated at the USC/Westside Cancer Center, USC/Norris Comprehensive Cancer Center, or LAC + USC Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2014-12-23 (Actual); Primary Completion 2016-06-08 (Actual); Study Completion 2016-06-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with elevated CTCs | Up to 2 years
  Descriptive statistics will also be applied to summarize levels of CTC numbers. The predominant statistical approaches will include correlation indices and mean comparisons to explore relations within the full data set and between clinical variables and expression data. The predominant statistical approaches will include correlation indices and mean comparisons to explore relations within the full data set and between clinical variables and expression data. The proportion of patients with elevated CTCs will be estimated using a 90% confidence interval.
Expression of individual markers according to clinical stage, serum PSA, and pathologic grade | Up to 2 years
  Descriptive statistics will also be applied to summarize expression of individual markers according to clinical variables (clinical stage, serum PSA, pathologic grade, etc). The predominant statistical approaches will include correlation indices and mean comparisons to explore relations within the full data set and between clinical variables and expression data.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Gross, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States